CLINICAL TRIAL: NCT06895785
Title: Exalt Single-use Duodenoscope Vs Reusable Scope, a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Neal Ambrish Mehta, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RUMC-ORA-24022203
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Biliary Diseases; Pancreatic Duct Disorder
Keywords: endoscopic retrograde cholangiopancreatography (ERCP); duodenoscope; single-use; reusable; biliary disorder; pancreatic duct disorder
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Exalt Model D (Experimental): Exalt Model D single use duodenoscope will be used for ERCP
  Interventions: Device: Exalt Model D
- Standard Reusable (Active Comparator): Standard reusable model of duodenoscope will be used for ERCP
  Interventions: Device: Reusable

INTERVENTIONS:
Device: Exalt Model D — Exalt Model D single-use duodenoscope will be used in ERCP
  Other Names: Single-use duodenoscope
  Arms: Exalt Model D
Device: Reusable — Standard reusable duodenoscope will be used in ERCP
  Arms: Standard Reusable

SUMMARY:
This randomized controlled trial (RCT) is designed to evaluate the new generation Exalt Model disposable duodenoscope compared to the reusable scope in terms of feasibility, ease of use, adverse events, number of crossover events, and infection rates.

DETAILED DESCRIPTION:
To ensure a safe and high-quality endoscopy, there are multiple disinfection protocols for endoscopes. Side-viewing duodenoscopes with an adjustable accessory device (elevator) contain potential blind spots for debris and bacteria that require specialized cleaning and disinfection methods beyond standard protocols for other endoscopes. It is thought that the duodenoscope's design, persistent postprocedural microbial contamination and biofilm formation make it more prone to cross-contamination5. Gromski et al, found there are documented pathogenic transmissions, which led to harm in multiple patients and centers3. Infection control was likely related to two major components, reusable duodenoscopes and procedural factors related to how the reusable duodenoscopes were reprocessed3. Multidrug-resistant organisms, such as carbapenem-resistant Enterobacteriaceae, that were associated with reusable duodenoscopes lead the FDA to mandate the transition to improved cleaning and disinfection methods or single-use platforms to eliminate infection transmission. One such single-use platform is the Exalt Model D (Boston Scientific, Marlboro, MA), which received FDA approval in 2020 for use of single-use duodenoscopes. Early iterations of the Exalt were used on a case-by-case basis per institution-specific protocols, mainly due to the learning curve involved with using the scope. A new version of Exalt has been released to market in 2023 with modifications that may make it more feasible to use in all settings requiring a duodenoscope. This randomized controlled trial (RCT) is designed to evaluate the new generation Exalt Model disposable duodenoscope compared to the reusable scope in terms of feasibility, ease of use, adverse events, number of crossover events, and infection rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18 years old who have biliary or pancreatic duct disorder, based on clinical symptoms and radiological findings at CT or magnetic resonance cholangiopancreatography
* Native papilla

Exclusion Criteria:

* Patients with altered pancreaticobiliary anatomy
* Pregnancy
* Patients with percutaneous transhepatic biliary drainage
* Prior history of ERCP
* Inability to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Number of attempts required to achieve successful cannulation of the desired duct | From the time of the ERCP to 7 days post-ERCP per standard of care
  Measure and compare the total number of attempts required to achieve successful cannulation of the desired duct.

SECONDARY OUTCOMES:
Crossover single to reusable | From the start of the ERCP to the end of procedure
  The incidence of crossovers from single-use duodenoscope to reusable duodenoscope
Use of advanced cannulation techniques | From the start of the ERCP to the end of procedure
  The utilization of advanced cannulation techniques in ERCP procedure
Performance on ERCP maneuvers | From the start of the ERCP to the end of procedure
  Subjective ratings on 14 ERCP maneuvers. ("not preferred/neutral/preferred" relative to the reusable duodenoscope endoscopist usually uses in clinical practice), 23 device performance characteristics. (Likert scale of 1 [not preferred] to 5 [comparable with reusable duodenoscope])
Adverse events | From the completion of the ERCP to 7 days post-ERCP per standard of care
  Post- ERCP pancreatitis, post-sphincterotomy bleed, and infection at 72 hours and 7 days post-ERCP procedure per Standard of Care.
Endoscopist-determined ease of use | From the start of the ERCP to the end of procedure
  Median overall satisfaction with the single-use duodenoscope during the procedure (Likert scale of 1 [unsatisfied] to 10 [very satisfied], followed by the option "If you answered ≤ 5, specify reason")

CONTACTS AND LOCATIONS:
Overall Officials: Neal A Mehta, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided